CLINICAL TRIAL: NCT01586091
Title: Comparison of Efficacy and Consistency of Action of Levocetirizine 5 mg Once Daily With Fexofenadine 60 mg Twice Daily in the Histamine Induced Wheal, Flare and Itch Response
Brief Title: Safety Study of Levocetirizine and Fexofenadine
Acronym: LAWAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Martin Metz, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-022747-38
Record Dates: First submitted 2012-04-23; First posted 2012-04-26 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Pruritus; Chronic Urticaria; Allergic Rhinitis
MeSH Terms: conditions — Pruritus; Chronic Urticaria; Rhinitis, Allergic | interventions — levocetirizine; fexofenadine; Tablets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo per os at time 0 hours + placebo per os at 12 hours.
  Interventions: Drug: Placebo Oral Tablet
- Levocetirizin (Active Comparator): Levocetirizin 5mg at time 0 and placebo per os at 12 hours
  Interventions: Drug: Levocetirizine Oral Tablet; Drug: Placebo Oral Tablet
- Fexofenadine (Active Comparator): Fexofenadine 60mg per os at time 0 hours + fexofenadine 60mg per os at 12 hours
  Interventions: Drug: Fexofenadine 60 Mg Oral Tablet

INTERVENTIONS:
Drug: Levocetirizine Oral Tablet
  Arms: Levocetirizin
Drug: Fexofenadine 60 Mg Oral Tablet
  Other Names: Telfast
  Arms: Fexofenadine
Drug: Placebo Oral Tablet
  Other Names: Lichtenstein
  Arms: Levocetirizin; Placebo

SUMMARY:
This Study is to comparison of Efficacy and Consistency of Action of Levocetirizine 5 mg once daily with Fexofenadine 60 mg twice daily in the histamine induced wheal, flare and itch Response.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled study with intra-individual comparison of the histamine induced wheal and flare reaction. In September 2009, Fexofenadine was approved as an antihistamine against allergies in Japan and it is currently used widely. It has been approved in 120 countries, including the US, UK, France and Germany [11]. In Europe and the United States, fexofenadine is marketed at 120 mg once daily for allergic rhinitis and 180mg once daily for urticaria. In Japan, fexofenadine is marketed at 60 mg twice daily for both conditions. But is this dosage regimen as effective as levocetirizine, 5 mg once daily? The above described study from Takahashi et al, comparing 60 mg twice daily versus cetirizine 10 mg once daily suggests that it is not [4]. The aim of the study is to compare the efficacy and consistency of action of levocetirizine 5 mg once daily with fexofenadine 60 mg twice daily over a 24 hour period in the histamine induced wheal, flare and itch response. Furthermore, we would like to investigate whether a different between Japanese and Caucasian exists or not. Each volunteer will receive the study medication at time point 0 and 12 hour later. Skin Prick Test (SPT) will be performed in each volunteer using histamine (10 mg/ml), 15 minutes before drug admission (baseline) and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours afterwards. Volumetric optical scanning system and infrared camera will be used for objective evaluation of the wheal- and flare reduction. Additionally, measurement of the erythema diameter with a transparent ruler will be performed. The subjective intensity of itching will be assessed using a Visual Analogue Scale (VAS). To relate the pharmacokinetics of the drugs to their pharmacodynamics, blood samples for assay of drug concentrations will be taken at baseline and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours later. Subjects will undergo the same procedure on three separate occasions to receive each treatment option. The options are: placebo at time 0 hours + placebo at 12 hours, Levocetirizine 5mg at time 0 hours + placebo at 12 hours or fexofenadine 60mg at time 0 hours + fexofenadine 60mg at 12 hours. There will be a washout period of at least 6 days between the treatments.

ELIGIBILITY:
Inclusion Criteria:

Eighteen (18) healthy male volunteers, including at least 6 persons of Japanese origin, will be recruited for this study

Exclusion Criteria:

* None of the subjects will have taken oral antihistamines, antidepressants, antipsychotics or corticosteroids or applied topical antihistamines, corticosteroids or mast cell stabilizers to the skin for 2 weeks prior to testing.
* No subject shall perform physical exercise for 4 hours prior to the skin prick testing.
* Especially, Bronchial asthma, anaphylactic reactions in the history, use of beta-blockers, skin diseases in the test field are exclusion criteria.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, MD, Principal Investigator — Charite Universitätsmedizin Berlin
Locations (1):
- University of Berlin Charité, Department of Dermatology and Allergy, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available.

REFERENCES:
- [Derived] Schoepke N, Church MK, Maurer M. The inhibition by levocetirizine and fexofenadine of the histamine-induced wheal and flare response in healthy Caucasian and Japanese volunteers. Acta Derm Venereol. 2013 May;93(3):286-93. doi: 10.2340/00015555-1490. PMID 23147964

RESULTS

PARTICIPANT FLOW:
Groups:
- Day 1: Intake of Placebo- Fexofenadine 6 mg - Levocetirizin 5 mg
- Day 2: Intake of Fexofenadine 6 mg - Levocetirizin 5 mg - Placebo
- Day 3: Intake of Placebo- Levocetirizin 5 mg- Fexofenadine 60
Period: Overall Study
Arm/Group | Day 1 | Day 2 | Day 3
Started | 6 (9 Caucasian and 9 Asian participants, each received Levocetiricine, fexofenadine and Placebo.) | 6 (9 Caucasian and 9 Asian participants, each received Levocetiricine, fexofenadine and Placebo.) | 6
Completed | 6 (9 Caucasian and 9 Asian participants, each received Levocetiricine, fexofenadine and Placebo.) | 6 (9 Caucasian and 9 Asian participants, each received Levocetiricine, fexofenadine and Placebo.) | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Day 2: Intake on 0 hours and 12 hours Intake Levocetirizn
- Day 3: Intake on 0 hours and 12 hours Intake Fexofenadine
- Day 1: Intake on 0 hours and 12 hours Intake Placebo
- Total: Total of all reporting groups
Arm/Group | Day 2 | Day 3 | Day 1 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: A total of 9 Patients (includes Asian and Caucasian) per Arm/Group were analysed.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 3 | 3 | 3 | 9
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 3 | 3 | 3 | 9
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Germany | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Pruritus as Assessed by the VAS Score
Description: We measured drug concentrations and various aspects of skin provocation testing such as itch intensity and wheal size. Measurements made at each time point were as followed: Pruritus was assessed every 30 s for 10 min after SPT using a visual analogue scale (VAS) score with a "0" and "100" at the two ex- tremes of an unmarked 100 mm line with higher values indicating greater puritus. The mean VAS for each 10 min was calculated and used as a primary end Point.
Time Frame: up to 10 minutes after skin prick test performed 24 hours after drug administration
Population: Please see Outcome Measure Description. Itch was measured using a 10 point VAS.
Measure: Mean (Standard Error); unit: mm
Groups:
- Levocetirizin: 5 mg once daily
- Fexofenadine: 60 mg twice daily
- Placebo: Placebo as comparison to Levocetirizin
Arm/Group | Levocetirizin | Fexofenadine | Placebo
Number analyzed (Participants) | 18 | 18 | 18
mm | 11.5 (16.4) | 25.4 (35.3) | 46.0 (44.6)

2. Primary Outcome: Flaire Diameter (mm)
Description: Flaire diameter was measured with a transparent ruler as the mean of the largest diameter and the diameter at right angles to this.
Time Frame: 24 hours per treatment
Population: Please see Outcome measure description. Flair Diameter was measured in mm.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Placebo | Levocetirizin | Fexofenadine
Number analyzed (Participants) | 18 | 18 | 18
mm | 69.4 (24.8) | 20.4 (10.0) | 39.9 (13.6)

3. Primary Outcome: Wheal Volume (cm3)
Description: Wheal volume was measured by a non-contact three dimensional measurement system (PRIMOS contact, GFM Messtechnik GmbH, Teltow, Germany).
Time Frame: 24 hours per treatment
Population: Please see Outcome Measure Description. Wheal volume was measured in cm3. The units of measure are provided in the report of the this study protocol.
Measure: Mean (Standard Error); unit: cm3
Arm/Group | Placebo | Levocetirizin | Fexofenadine
Number analyzed (Participants) | 18 | 18 | 18
cm3 | 174.6 (50.9) | 35.2 (13.5) | 106.3 (39.5)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected on the following time points: 0 (baseline), 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours
Groups:
- Levocetirizine: 5 mg once daily
- Fexofenadine: 60 mg twice daily, oral
- Placebo: Placebo against Levocetirzine
Arm/Group | Levocetirizine | Fexofenadine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/18 | 3/18 | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levocetirizine (N=18) | Fexofenadine (N=18) | Placebo (N=18)
fatigue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
pain at the puncture site of the intravenous catheter (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
bacterial inflammation of the finger (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
pain in the knee joint (Social circumstances) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes